CLINICAL TRIAL: NCT06115655
Title: A Single-center, Prospective Cohort Study on the Differentiation of Benign and Malignant Bile Duct Stenosis Based on Bile and Peripheral Blood cfDNA Methylation Profiles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Other Study IDs: KY20232312
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Bile Duct Neoplasms; Jaundice, Obstructive; Bile Duct Diseases
Keywords: Methylation; Liquid Biopsy; Cell-Free Nucleic Acids; Cancer Diagnosis
MeSH Terms: conditions — Bile Duct Neoplasms; Jaundice, Obstructive; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml peripheral venous blood sample and 5ml bile from each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- malignant patients: The presence of biliary stricture due to malignant diseases, such as cholangiocarcinoma.
  Interventions: Diagnostic Test: cfDNA methylation detection
- benign patients: The presence of biliary stricture due to benign diseases, such as inflammation.
  Interventions: Diagnostic Test: cfDNA methylation detection

INTERVENTIONS:
Diagnostic Test: cfDNA methylation detection — Extract cfDNA from bile and plasma, and perform methylation detection.

SUMMARY:
The goal of this observational study is to detect the methylation characteristics of cfDNA in the bile and plasma of patients with bile duct stricture. The main question it aims to answer is: Can the developed model, using peripheral blood and bile cell-free DNA sequencing, work well in screening and classifying unknown biliary stricture? Participants will collect approximately 10ml of peripheral blood and 5ml of bile from the patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with biliary stricture aged between 18 and 90 years old.
* 2. Patients scheduled to undergo ERCP surgery due to obstructive jaundice or cholangitis.
* 3. Definite benign or malignant diagnosis: with a pathological diagnosis of benign or malignant disease, or with follow-up data indicating a benign or malignant diagnosis.

Exclusion Criteria:

* 1. Receive radiotherapy, chemotherapy, or targeted therapy before sampling.
* 2. Malignant tumors in other parts of the body (not related to biliary stricture).
* 3. Unable to determine the nature of the biliary stricture.
* 4. Ineligible for ERCP due to systemic conditions or gastrointestinal obstruction.
* 5. Pregnant or breastfeeding women.
* 6. Unable to sign the informed consent form.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the "Sample Size Calculation for Comparative Diagnostic Studies with Categorical Variables (Rates)" method, it is calculated. Based on the previous research results, it is estimated that the diagnostic sensitivity of sequencing methylation profiles in bile cfDNA is 82%, the specificity is 95%, the allowable error in sensitivity is 0.1, the allowable error in specificity is 0.1, α is set to 0.05, the loss to follow-up rate is 10%, and the calculated sample size is approximately 161 cases.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | Immediately after test completion
  This refers to the ability of the test (cell-free DNA sequencing) to correctly classify individuals into the categories of having or not having the disease. It is a measure of the test's overall effectiveness. The reference test is histological test for cancers or one-year follow-up for non-cancers.
Sensitivity | Immediately after test completion
  This is the ability of the test (cell-free DNA sequencing) to correctly identify those with the disease. It is the proportion of true positive results (those with the disease who test positive) to the total number of individuals who actually have the disease. The reference test is histological test for cancers or one-year follow-up for non-cancers.
Specificity | Immediately after test completion
  This is the ability of the test (cell-free DNA sequencing) to correctly identify those without disease. It is the proportion of true negative results (those without the disease who test negative) to the total number of individuals who actually do not have the disease. The reference test is histological test for cancers or one-year follow-up for non-cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — The First Affiliated Hospital of the Air Force Medical University
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorrell R, Pawa S, Zhou Y, Lalwani N, Pawa R. The Diagnostic Dilemma of Malignant Biliary Strictures. Diagnostics (Basel). 2020 May 25;10(5):337. doi: 10.3390/diagnostics10050337. PMID 32466095
- [Background] Dumonceau JM, Delhaye M, Charette N, Farina A. Challenging biliary strictures: pathophysiological features, differential diagnosis, diagnostic algorithms, and new clinically relevant biomarkers - part 1. Therap Adv Gastroenterol. 2020 Jun 16;13:1756284820927292. doi: 10.1177/1756284820927292. eCollection 2020. PMID 32595761
- [Background] Sun B, Moon JH, Cai Q, Rerknimitr R, Ma S, Lakhtakia S, Ryozawa S, Kutsumi H, Yasuda I, Shiomi H, Li X, Li W, Zhang X, Itoi T, Wang HP, Qian D, Wong Lau JY, Yang Z, Ji M, Hu B; Asia-Pacific ERCP Club. Review article: Asia-Pacific consensus recommendations on endoscopic tissue acquisition for biliary strictures. Aliment Pharmacol Ther. 2018 Jul;48(2):138-151. doi: 10.1111/apt.14811. Epub 2018 Jun 7. PMID 29876948
- [Background] Davalos V, Esteller M. Cancer epigenetics in clinical practice. CA Cancer J Clin. 2023 Jul-Aug;73(4):376-424. doi: 10.3322/caac.21765. Epub 2022 Dec 13. PMID 36512337
- [Background] Vedeld HM, Grimsrud MM, Andresen K, Pharo HD, von Seth E, Karlsen TH, Honne H, Paulsen V, Farkkila MA, Bergquist A, Jeanmougin M, Aabakken L, Boberg KM, Folseraas T, Lind GE. Early and accurate detection of cholangiocarcinoma in patients with primary sclerosing cholangitis by methylation markers in bile. Hepatology. 2022 Jan;75(1):59-73. doi: 10.1002/hep.32125. Epub 2021 Dec 5. PMID 34435693
- [Background] Goeppert B, Stichel D, Toth R, Fritzsche S, Loeffler MA, Schlitter AM, Neumann O, Assenov Y, Vogel MN, Mehrabi A, Hoffmann K, Kohler B, Springfeld C, Weichenhan D, Plass C, Esposito I, Schirmacher P, von Deimling A, Roessler S. Integrative analysis reveals early and distinct genetic and epigenetic changes in intraductal papillary and tubulopapillary cholangiocarcinogenesis. Gut. 2022 Feb;71(2):391-401. doi: 10.1136/gutjnl-2020-322983. Epub 2021 Jan 19. PMID 33468537
- [Background] Colyn L, Barcena-Varela M, Alvarez-Sola G, Latasa MU, Uriarte I, Santamaria E, Herranz JM, Santos-Laso A, Arechederra M, Ruiz de Gauna M, Aspichueta P, Canale M, Casadei-Gardini A, Francesconi M, Carotti S, Morini S, Nelson LJ, Iraburu MJ, Chen C, Sangro B, Marin JJG, Martinez-Chantar ML, Banales JM, Arnes-Benito R, Huch M, Patino JM, Dar AA, Nosrati M, Oyarzabal J, Prosper F, Urman J, Cubero FJ, Trautwein C, Berasain C, Fernandez-Barrena MG, Avila MA. Dual Targeting of G9a and DNA Methyltransferase-1 for the Treatment of Experimental Cholangiocarcinoma. Hepatology. 2021 Jun;73(6):2380-2396. doi: 10.1002/hep.31642. PMID 33222246